CLINICAL TRIAL: NCT03566329
Title: Control of Emergence Hypertension After Craniotomy: Comparison Between the Efficacy of Magnesium Sulphate and Lidocaine Infusion (Randomized Controlled Study)
Brief Title: Magnesium Sulphate Versus Lidocaine for Control of Emergence Hypertension
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed Mohamed ELbadawy (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed ELbadawy, Ahmed Mohamed ELbadawy- Clinical investigator , Cairo University, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N2011
Record Dates: First submitted 2018-06-10; First posted 2018-06-25 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Craniotomy; Hypertension
Keywords: craniotomy- Emergence- hypertension
MeSH Terms: conditions — Hypertension | interventions — Magnesium Sulfate; Lidocaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Magnesium sulphate (Active Comparator): 50 mg/kg over 10 minutes loading followed by 15mg/kg/hr infusion
  Interventions: Drug: Magnesium sulphate
- lidocaine hydrochloride (Active Comparator): 1.5mg/kg loading followed by 2mg/kg/hr infusion
  Interventions: Drug: Lidocaine Hydrochloride
- NaCl 0.9% normal saline (Placebo Comparator): Normal saline infusion with the same rate as the study drugs
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Magnesium sulphate — Magnesium sulphate 50 mg/kg over 10 minutes loading followed by 15mg/kg/hr infusion. .
  Arms: Magnesium sulphate
Drug: Lidocaine Hydrochloride — lidocaine hydrochloride 1.5mg/kg loading followed by 2mg/kg/hr infusion
  Other Names: Xylocaine
  Arms: lidocaine hydrochloride
Drug: Normal saline — Normal saline infusion with the same rate of infusion as the study drugs
  Other Names: Nacl
  Arms: NaCl 0.9% normal saline

SUMMARY:
Post-craniotomy emergence hypertension is a common phenomenon that may predispose to development of intracranial hematoma and cerebral edema.The aim of this study is to compare the safety and efficacy of Mgso4 versus lidocaine infusion for control of emergence hypertension after craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status Ι or Π.
* scheduled patients for brain tumor excision.

Exclusion Criteria:

* Hepatic, renal, cardiac, pulmonary, or endocrine impairment.
* Signs of increased intracranial pressure or allergy to any of the used drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
postcraniotomy emergence hypertension response to the study drugs | 4hours
  The number of the patients who have systolic blood pressure below 140 mmH during emergence of anesthesia after craniotomy for brain tumors in each group

SECONDARY OUTCOMES:
Recovery time | 2 hours
  Time till discharge from PACU
Incidence of side effects of the used drugs | 4 hours
  measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed ELbadawy, MD, Principal Investigator — Faculty of medicine- Cairo University- Egypt
Locations (1):
- Ahmed ELbadawy, Cairo, Egypt